CLINICAL TRIAL: NCT06535373
Title: Restrict and Strengthen: Unraveling the Impact of Blood Flow Restriction Training on Upper Extremity Grip Strength
Brief Title: Blood Flow Restriction Training on Upper Extremity Grip Strength
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Casa Colina Hospital and Centers for Healthcare (Other)
Collaborators: Azusa Pacific University (Other)
Responsible Party: Principal Investigator, Emily Rosario, DIrector of Research, Casa Colina Hospital and Centers for Healthcare
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BFRGRIP
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled study where participants will be randomly assigned to one of two groups.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood flow restriction with low-weight resistance training (LWRT) group (Experimental): a blood flow restriction with low-weight resistance training (LWRT) group
  Interventions: Other: Blood flow restriction
- No Blood flow restriction group which just does LWRT (No Intervention): a non blood flow restriction group which just does low-weight resistance training

INTERVENTIONS:
Other: Blood flow restriction — Both groups will undergo a 6-week training intervention with training 2x a week, after which grip strength and other relevant outcomes will be measured and compared. Exercise sessions will be at least 48 hours apart. Participants will be allowed to continue with their normal exercise routine outside of the study.
  Arms: Blood flow restriction with low-weight resistance training (LWRT) group

SUMMARY:
The primary objective of this prospective study is to investigate the effects of Blood Flow Restriction (BFR) training compared to traditional low-weight resistance training on grip strength in young adults.

Despite the growing interest in BFR training and its potential benefits, there is limited research specifically investigating its impact on grip strength. Understanding the effects of BFR training on grip strength could have significant implications for individuals seeking to optimize their grip performance, rehabilitation settings, and sports performance enhancement. Additionally, examining the safety and efficacy of BFR training for this specific outcome will contribute valuable insights to the scientific community.

DETAILED DESCRIPTION:
Blood Flow Restriction (BFR) training, also known as occlusion training, is an innovative exercise technique that involves using a tourniquet or blood pressure cuff to partially restrict blood flow to the working muscles during resistance exercises. This unique approach allows individuals to achieve significant muscle strength and hypertrophy gains with lower resistance loads, making it a promising alternative to traditional high-intensity training methods. BFR training has been extensively studied in various populations, demonstrating its potential benefits for muscle growth, strength, and endurance across different muscle groups.

While much research has focused on the effects of BFR training on large muscle groups like the quadriceps and biceps, there is a paucity of studies specifically investigating its impact on upper extremity grip strength. Grip strength is a fundamental measure of hand and forearm muscle function, playing a crucial role in various activities of daily living, occupational tasks, and sports performance. Understanding the effects of BFR training on grip strength could provide valuable insights into optimizing hand and forearm strength and functional capacity.

The current study seeks to fill this research gap by examining the effects of Blood Flow Restriction (BFR) training on upper extremity grip strength in a healthy young adult population. By exploring this novel application of BFR training, we aim to contribute to the existing body of knowledge surrounding BFR's potential benefits for grip strength enhancement. The results of this study may have implications for athletes, rehabilitation programs, and individuals seeking efficient and effective ways to enhance their grip strength and overall upper extremity function.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between 18 and 35 years old at the time of enrollment.

Participants should be in good general health with no known cardiovascular, musculoskeletal, or neurological disorders that could interfere with exercise participation.

Participants must provide informed consent before enrollment in the study, indicating their willingness to participate voluntarily.

Exclusion Criteria:

* Participants with a history of cardiovascular disease (e.g., heart disease, hypertension), musculoskeletal injuries (e.g., fractures, dislocations), or neurological disorders (e.g., neuropathy) that could affect exercise performance will be excluded.

Participants taking medications or supplements that may impact muscle strength, metabolism, or blood flow will be excluded from the study.

Pregnant individuals will be excluded due to potential risks associated with exercise and blood flow restriction during pregnancy.

Individuals with recent upper extremity injuries, such as strains, sprains, or fractures, will be excluded until fully recovered.

Blood Pressure: Participants with uncontrolled high blood pressure or other medical conditions affecting vascular health may be excluded due to potential risks associated with blood flow restriction.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Grip Strength | baseline, post-intervention (6 weeks), and follow-up (6 weeks)
  Isometric grip strength will be assessed in the dominant arm after the intervention using the Jamar hydraulic hand dynamometer (Lafayette Instruments, Lafayette, IN). Participants will be positioned in sitting with the knees and hips flexed to 90 degrees and feet flat on the floor. The shoulder will be in a neutral position with the elbow flexed to 90 degrees and the forearm in neutral pronation-supination. (Crotin & Ramsey, 2021) The participant will be instructed to squeeze the dynamometer with maximal effort for 3 seconds while receiving verbal encouragement. A total of three repetitions will be completed with a 30 second rest between trials to reduce fatigue. (Crotin & Ramsey, 2021) The peak grip strength value of all three trails will be used for baseline strength and 30% of the peak value will be used to calculate the resistance (in lbs.) for the exercise protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Casa Colina Healthcare and Hospital, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: Undecided